CLINICAL TRIAL: NCT00481819
Title: A Multicenter, Randomized, Open Label, Parallel Study to Evaluate and Compare the Efficacy and Safety of FK506MR vs Prograf® in Combination With MMF and Steroids in Patients Undergoing Kidney Transplantation and a Pharmacokinetics Study.
Brief Title: A Study to Compare the Efficacy and Safety of FK506MR vs Prograf® in Patients Undergoing Kidney Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MR4KTxCN01
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Tacrolimus; Methylprednisolone; Prednisolone; Mycophenolate Mofetil
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Methylprednisolone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): In combination with MMF and steroids
  Interventions: Drug: FK506MR; Drug: Mycophenolate Mofetil; Drug: Methylprednisolone; Drug: Prednisolone
- 2 (Active Comparator): In combination with MMF and steroids
  Interventions: Drug: Prograf; Drug: Mycophenolate Mofetil; Drug: Methylprednisolone; Drug: Prednisolone

INTERVENTIONS:
Drug: FK506MR — oral
  Other Names: Advagraf; Tacrolimus modified-release; MR4
  Arms: 1
Drug: Prograf — oral
  Other Names: tacrolimus; FK506
  Arms: 2
Drug: Mycophenolate Mofetil — oral
  Other Names: MMF
Drug: Methylprednisolone — oral
Drug: Prednisolone — oral

SUMMARY:
The patients about to undergo kidney transplantation will be randomized to one of the following two group:

Group FK506MR: FK506MR/MMF/steroid; Group Prograf® : Prograf® /MMF/steroid. The treatment period is 3 months( 12 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent with the date of the patient must be obtained.
* Patient between 18-70 years of age receiving the primary kidney.
* Female patients must have a negative pregnancy test prior to the enrolment.
* Female patients of child bearing potential must agree to practice effective birth control during the study.

Exclusion Criteria:

* Kidney re-transplantation patients or received an organ transplantation other than a kidney.
* PRA>10% in the previous 6 months.
* Patient who need antibody induction therapy.
* Patient with significant liver disease, defined as having continuously elevated >2 times of SGPT and/or SGOT and/or total bilirubin levels during the past 28 days.
* Patient with severe infection requiring treatment, and/or severe diarrhea, vomiting, active upper gastrointestinal tract malabsorption or active peptic ulcer.
* Patient has any history of severe cardiovascular, respiratory disease; or history of malignancy.
* Patient is HIV or HBsAg positive.
* Patient is allergic to Prograf or macrolide antibiotics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Event rate of patients with acute rejections | 12 weeks

SECONDARY OUTCOMES:
Incidence of and time to acute rejections | 12 Weeks
Overall frequency of acute rejections | 12 Weeks
Rate of patient and graft survival following transplantation | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Ao Jianhua, Principal Investigator — Department of Urologic Surgery
Locations (9):
- China (9):
  - 3 Sites, Beijing, Beijing Municipality
  - Fuzhou, Fujian
  - 2 Sites, Guangzhou, Guangdong
  - Wuhan, Hubei
  - Changsha, Hunan
  - Shenyang, Liaoning
  - 2 Sites, Shanghai, Shanghai Municipality
  - Chongqing, Sichuan
  - Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided